CLINICAL TRIAL: NCT05764512
Title: Endorphins Applied to Women Who Have Delivered Vaginally Effect of Massage on Pain
Brief Title: Endorphin Massage Application to Women Who Gave Birth Vaginally
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nurseli Soylu Erener, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023/09
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Pain; Birth, First
Keywords: Birth; Vaginal Birth; Massage; Pain; Endorphin
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Two gruops with intervention gruop and control grup.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The blood samples are numbered by writing the names of the puerperant women. Nurses who care, the biochemist who analyzes the blood samples and the specialist who does the statistical analysis will not know the groups to which the puerperal puerperants are assigned. In the hospital where the research will be conducted, one of the two parts of the postpartum service is used for the intervention group and the other for the control group in order to prevent encounters between the intervention and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Is the group to which endorphin massage will be applied. Endorphin massage is a gentle touch and massage method that can improve the relaxation state in the body through the skin surface.
  Interventions: Other: Endorphin massage
- Control gruop (No Intervention): No application will be made.

INTERVENTIONS:
Other: Endorphin massage — With the anterior surface of the fingertips of the hand, a "V" will be drawn slowly, starting from the sacral region and towards the ribs. The same process will be continued from the sacral region until the 7th cervical vertebra.
  From the 7th cervical vertebra, the front surface of the fingertips will be descended first to the shoulders and then to the dorsal region of the upper and forearms in turn.
  Starting from the dorsal region of the forearm, the first stage of the massage will end by descending to the upper arm, shoulders, 7th cervical vertebra, spine and sacral region with the back of the thumbs. These massage steps will be repeated until 20 minutes are completed.
  Endorphin massage will be applied every 2 hours.
  Arms: Intervention group

SUMMARY:
In this study, it is aimed to determine the effect of endorphin massage applied to puerperant women who had vaginal delivery on pain, comfort, mood and serum beta endorphin levels in the postpartum period.

DETAILED DESCRIPTION:
Massage application provides an increase in the level of endorphins by making a relaxing effect on the muscles. Endorphin massage increases the release of endorphins, allowing the individual to relax, relax the muscles and reduce pain. Endorphin massage is a light massage technique that can increase the release of oxytocin and endorphin hormones, providing a feeling of calmness and comfort. In addition to reducing pain, the endorphin hormone provides relaxation, supports the immune system, and accelerates metabolic activities. It is also known as the happiness hormone.

It is stated that back massage will increase the release of endorphin hormones by relaxing the mother. In other studies conducted in the postpartum period, it has been determined that massage applied reduces the severity of pain and stress, and increases the level of comfort.

Studies have shown that endorphin massage applied to pregnant women reduces back pain. In another study, it was determined that deep tissue massage applied to the back area after cesarean section reduced the level of pain. In the other study, it was determined that the endorphin massage applied to the 3rd trimester pregnant women reduced the level of anxiety.

When the literature is examined, no study has been found that examines the effect of endorphin massage applied to puerperant women on pain, comfort, mood and beta endorphin levels in the postpartum period. The fact that endorphin massage is applied to similar areas with both back massage and oxytocin massage suggests that endorphin massage may affect the pain process experienced in the postpartum period. It is aimed to determine the effect on endorphin level.

ELIGIBILITY:
Inclusion Criteria:

* 37-40. Those who gave birth vaginally in their gestational week,
* In the first 24 hours postpartum,
* Primiparous,
* Episiotomy applied,
* Having a VAS value of at least 5 points,
* Having given birth to a single baby,
* Your baby's APGAR Score is between 7-10,
* Skin-tissue integrity,
* No communication problem,
* The spoken language is Turkish,
* Voluntary to participate in the study

Exclusion Criteria:

* The baby was admitted to the neonatal intensive care unit,
* Having a cesarean section,
* Experiencing risky labor,
* Postpartum bleeding,
* Epidural analgesia applied
* Having a psychiatric disease (Bipolar Disorder, Depression, Obsessive Compulsive Disorder),
* Having chronic disease (Heart disease, Thyroid problems, Diabetes mellitus, Hypertension, asthma, COPD),
* Postpartum women diagnosed with risky pregnancy (Pre-eclampsia, Eclampsi, Pregnancy-related hypertension, Gestational diabetes, bleeding conditions during pregnancy)

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | two hours
  It is a commonly used scale to measure pain. It consists of a 10 cm ruler on which the patient marks the pain, showing that there is no pain at one end and unbearable pain at the other end. The distance between the point where the patient marked the pain and the pain-free interval is measured in cm and recorded.
  In addition, this scale is used to measure comfort. The VAS, which will be used to determine the level of comfort, consists of a ruler of 0 to 10 cm, as well as the level of pain. VAS; 0 = very comfortable, 10 = extremely uncomfortable. In the calculation of the comfort score, the distance between the place marked by the puerperant as "I am comfortable" and the place marked as "I am uncomfortable" is measured and recorded in cm. In this research, the Visual Analog Scale is used to measure both pain level and comfort level.
Brief Mood Introspection Scale | two hours
  In the 16-item scale, the items consist of the emotion adjective and aim to evaluate the current emotional state of the participants. By obtaining two types of scores with the scale, positive (8 items) and negative (8 items) mood levels of the participants are determined. High scores for both mood states indicate high positive or negative emotions. The highest score for both moods is 32 and the lowest score is 8.
Serum Beta Endorphin Level | two hours
  Blood samples are taken from the puerperal women by following the antiseptic rules, into a yellow-capped and gelled blood tube (3-4 mL) by the researcher. The blood tubes are kept at room temperature and in an upright position for 30 minutes. Samples sent to the laboratory are centrifuged at 4000 rpm for 10 minutes. The serum obtained after centrifugation is taken from the blood tubes, put into eppendorf tubes and stored frozen at -80 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Nurseli SOYLU ERENER, Principal Investigator — TC Erciyes University
Locations (1):
- Kayseri City Hospital, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Do not share until the article is published.

REFERENCES:
- [Background] Guney E, Ucar T. Effects of deep tissue massage on pain and comfort after cesarean: A randomized controlled trial. Complement Ther Clin Pract. 2021 May;43:101320. doi: 10.1016/j.ctcp.2021.101320. Epub 2021 Jan 28. PMID 33548749